CLINICAL TRIAL: NCT03399968
Title: Extracorporeal Shockwave Therapy (ESWT) in Patients Suffering From Complete Paraplegia at the Thoracic Level
Brief Title: Extracorporeal Shockwave Therapy (ESWT) to Improve Function in Chronic ASIA-A Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AUVA Trauma Center Meidling (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESWT_SCI/1.9-2014
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries
Keywords: shockwave; ESWT
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled double blinded clinical intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Experimental): Application of shockwaves non-invasively at the level of injury
  Interventions: Device: ESWT
- Placebo ESWT (Placebo Comparator): Positioning of the therapy head at the injury level without application of shockwaves
  Interventions: Device: Placebo ESWT

INTERVENTIONS:
Device: ESWT — at low energy, shockwaves are applied non-invasively at the injury level and 5 segments up and down of the spinal cord paravertebrally left and right
  Other Names: Extracorporeal shockwave therapy
  Arms: ESWT
Device: Placebo ESWT — the ESWT therapy head is positioned at the level of injury and is moved up and down identically as described in the Verum intervention group (ESWT) but without application of shockwaves. The sound which is normally produced by shockwave generation is played by high quality sound recordings in the same amount as in the Verum group
  Arms: Placebo ESWT

SUMMARY:
The global prevalence of spinal cord injury is estimated between 236 to 4187/Million. A spontaneous recovery of the sense-motoric function is decreasing with the time after injury and is only seen sporadically after 1 to 2 years. Treatment options are mainly limited to improvement of the quality of life.

The present prospective randomized study is intended as a double-blind, placebo controlled multi-center investigation. Patients suffering from chronic paraplegia (lesion between THII and THX, ASIA A = complete central lesion) at least for 1 year after the initial trauma without spontaneous remission of the last 6 months are considered to be included in the study. Meeting the inclusion criteria and signing the informed consent, patients are treated in one of the two study centers. At study inclusion, a baseline evaluation comprising neurological, neurophysiological, functional and clinical investigation is performed. Patients dedicated to the ESWT intervention group will be treated once a week over 6 weeks with local non-invasive low energy extracorporeal shockwave therapy (=6 treatments with an electrohydraulic device). The follow-up will include neurological, neurophysiological, clinical as well as functional evaluation at the time points 6 weeks, 3 months and 6 months. Additionally, patients will be provided with a diary for documentation of drug adaptation, grade of spasticity and pain. Those patients dedicated to the Placebo ESWT group, will receive the identical scheme in treatment (but without application of shockwaves) and follow-up as the patients in the ESWT group. However, after positive completion of the study, these patients will be offered ESWT as well.

ELIGIBILITY:
Inclusion Criteria:

* patients with a spinal cord injury classified as ASIA A between the level of THII to THX (complete central lesion)
* at least 1 year after trauma
* no signs of spontaneous recovery over the last 6 months
* signed informed consent

Exclusion Criteria:

* central therapies over the last 6 months (eg stem cells, electro-therapy)
* Baclofen pump
* Joint contraction lower limb > 40° (hip or knee)
* Body weight > 135 kg
* Body height > 202 cm
* non-compliant patients
* Decubital ulcers at grade II or higher
* participation in an other clinical trial within the last 6 months
* Co-morbidities which make study completion doubtful or impossible
* Additional neurological diseases which may lead to further damage to the nerval system
* Malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-03-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Motor function | 24 weeks
  Motor function of the lower limbs assessed by gait analysis tool (Lokomat (R))

SECONDARY OUTCOMES:
Sensitivity and Motor function | 24 weeks
  Assessment of levels by the ASIA score ASIA score - a neurologic assessment for patients with spinal cord injury developed by the American Spinal Injury Association.
  Examination includes the pin-prick discrimination assessment at 28 specific sensory locations bilaterally but also 10 muscles bilaterally.
  Sensory levels for each dermatome (nt...not testable, 0...absent sensation, 1...present sensation but impaired, 2...normal) Motor function of 5 upper extremity and 5 lower extremity key muscles (0...complete paralysis, 1...palpable or visible contraction, 2...active movement, full range of motion, gravity eliminated, 3...active movement, full range of motion, against gravity, 4...active movement, full range of motion, against gravity and provides some resistance, 5...active movement, full range of motion, against gravity and provides normal resistance, nt...not testable)
Spasticity | 24 weeks
  Evaluation of spasticity degree assessed by the Tardieu test (muscle resistance to passive movement at both slow and fast speed) 2 measurements are performed:
  1. Quality of muscle reaction
  2. Angle of muscle reaction 3 speed definitions:
  1) V1 is slow as possible 2) V2 speed of limb falling under gravity 3) V3 moving as fast as possible Quality of Muscle Reaction (scored 0-5); 0 is no resistance to passive ROM to 5 indicating joint is immobile (Some versions scored 0-4).
Trunk control | 24 weeks
  evaluation of trunk control by the modified functional reach test and Ott test
Lung function | 24 weeks
  Assessment of lung function by peak flow measurements
Quality of life | 24 weeks
  Assessed by the disability scale SCIM (spinal cord independence measure); Subscores include self-care (range von 0-20 points), respiration and sphincter management (range from 0-40), and mobility (range from 0-40); In total scale range from 0-100 (0 = total dependence, 100 = complete independence).

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - AUVA Rehabilitation Center Weisser Hof, Klosterneuburg, Lower Austria
  - AUVA Rehabilitation Center Tobelbad, Haselsdorf, Styria

IPD SHARING:
Plan to Share IPD: No